CLINICAL TRIAL: NCT06275360
Title: Repositioning Immunotherapy in Veterans With Lung Cancer
Brief Title: Repositioning Immunotherapy in VetArans With Lung Cancer
Acronym: RIVAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPLP-002-23F
Record Dates: First submitted 2024-01-30; First posted 2024-02-23 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Carboplatin, paclitaxel, and nivolumab for three cycles followed by radiotherapy followed by nivolumab (for squamous cell lung cancer) OR Carboplatin, pemetrexed, and nivolumab for three cycles followed by radiotherapy followed by nivolumab (for lung adenocarcinoma)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Chemoimmunotherapy followed by radiotherapy (Experimental): Nivolumab (Opdivo) + plus platinum-doublet chemotherapy followed by radiotherapy
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Carboplatin, paclitaxel, and nivolumab for three cycles (for squamous cell lung cancer) or Carboplatin, pemetrexed, and nivolumab for three cycles (for lung adenocarcinoma) Followed by radiotherapy (60 Gy in 30 fractions) Followed by adjuvant nivolumab (six cycles)
  Other Names: Opdivo

SUMMARY:
This study is a multicenter Phase II single arm trial to assess the safety and efficacy of chemotherapy and immunotherapy followed by radiotherapy in patients with unresectable Stage III NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be more than 18 years of age.
* Patient must have a performance status of 0-1 (ECOG Performance Scale).
* Patient must be a candidate for concurrent chemoradiation.
* Unresectable Stage III NSCLC as assessed by investigator or multidisciplinary tumor board assessment
* PD-L1 tumor expression greater than or equal to 1%
* Presence of measurable disease according to RECIST v1.1
* Adequate organ function
* Available tissue (archival FFPE preferred) with adequate tumor content ( 20% tumor cellularity).

Exclusion Criteria:

* Active autoimmune disease that has requires immunosuppressive therapy in the previous year.
* Uncontrolled primary or acquired immunodeficiency (including HIV)
* Baseline corticosteroid usage (>10 mg prednisone or equivalent daily) aside from supportive medication use.
* Tumor with known EGFR, ALK, ROS1, MET or RET mutations/fusions.
* Presence of significant comorbidities precluding participation in a clinical study as determined by investigator.
* Prior thoracic radiotherapy or prior systemic treatment for stage IIIB/IV NSCLC
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with informed consent through 180 days after the last dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Has known active Hepatitis B or Hepatitis C.
* Has received a live vaccine within 30 days of enrollment.
* Known diagnosis of Interstitial Lung Disease
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Approximately two years after enrollment
  Defined as the time from start of treatment to radiographic/clinical progression (per irRECIST1.1), or death from any cause, whichever occurs first.
Treatment Tolerance | Approximately three years after enrollment
  Proportion of patients able to complete prescribed treatment course (all planned cycles of systemic therapy and all fractions of radiotherapy).

SECONDARY OUTCOMES:
Adverse Events | Approximately two years after enrollment
  Frequency of adverse events assessed by Common Terminology Criteria for Adverse Events (CTCAE) criteria 5.0 classified by body system, grade, and attribution.
Best overall response rate (BOR) | Approximately two years after enrollment
  Defined as the proportion of participants who achieve a confirmed either a best response of complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by central review.
Overall survival | Approximately two years after enrollment
  Defined as the time from start of treatment to the date of death from any cause..

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Green, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Nithya Ramnath, MD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (7):
- United States (7):
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No